CLINICAL TRIAL: NCT07037719
Title: Automatic Detection of Eligible Patients to RAUC Protocol (RAUCISABLE): a Retrospective Monocentric Pilot Study on Big-data
Brief Title: Automatic Detection of Eligible Patients to RAUC Protocol (RAUCISABLE)
Acronym: RAUCISABLE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2025_843_0015
Record Dates: First submitted 2025-06-11; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Emergency Department Visit
Keywords: Personalized medicine; augmented rehabilitation; artificial intelligence; emergency surgery; digestive surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients attending CHU Amiens-Picardie Emergency Department: Adults (age 17+), all ED patients

SUMMARY:
The augmented rehabilitation of emergency surgeries (ARES, RAUC in French) is a research program supported by Amiens-Picardy University Hospital and the University of Picardy Jules Verne. The RAUC program aims to enhance by multiple levers (enhanced recovery programs, artificial intelligence, organizational optimization, connected devices) the management of patients operated for digestive emergency surgery. RAUCisable aims to optimize the inclusion of eligible patients in the RAUC-AMIENS study and improve predictive models for patient management.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 17+), all ED patients

Exclusion Criteria:

* Patients who object to data use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending CHU Amiens-Picardie Emergency Department (ED).
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-01-17 (Estimated); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
Area Under the ROC Curve | 30 days
  Area Under the ROC Curve (AUROC) for RAUC-AMIENS inclusion

SECONDARY OUTCOMES:
AUROC and Mean Absolute Error | 30 days
  AUROC and Mean Absolute Error for continuous prediction of post-surgery LOS.
AUROC of unattended readmission | 30 days
  AUROC of unattended readmission
mean absolute error for readmission prediction | 30 days
  mean absolute error for readmission prediction

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc REGIMBEAU, MD, Principal Investigator — CHU Amiens-Picardie
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: Undecided